CLINICAL TRIAL: NCT05971953
Title: Effect of Muscle Energy Technique on Hamstring Muscle for the Trigger Points of Muscle of Mastication
Brief Title: Muscle Energy Technique on Hamstring Muscle for Trigger Points of Muscle of Mastication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01649Naureena Binte Sayed
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Trigger Point Pain, Myofascial; Temporomandibular Disorder
Keywords: trigger points; muscles of mastication; hamstring
MeSH Terms: conditions — Myofascial Pain Syndromes; Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Active Comparator): Muscle Energy Technique
  Interventions: Other: Muscle Energy Technique
- Conventional PT (Other): Hot pack Ischemic compression
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: Muscle Energy Technique — They would be receiving treatment as follow:
  The patient is instructed to gently attempt to push down on the practitioner's shoulder with the leg against the practitioner's resistance( 75% of his and her available strength). After the relaxation, the muscle is lengthened more aggressively beyond the barrier and held for up to 15 seconds. Frequency: 10 reps for 4 times/week for 2 consecutive weeks. Intensity: moderate intensity (pain free) Time: 20 mins
  Arms: Muscle Energy Technique
Other: Conventional PT — They would be receiving conventional treatment as follow:
  including hot pack for 10 mins ischemic compression for 60 seconds .Frequency: 5 reps with 60 sec hold for 4 times/week for 2 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 mins
  Arms: Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to find the effect of muscle energy technique for trigger points of muscle of mastication for reducing pain , improving mouth opening and jaw functional limitations.

DETAILED DESCRIPTION:
The primary muscles of mastication (chewing food) are the temporalis, medial pterygoid, lateral pterygoid, and masseter muscles. The masticatory muscles are divided into elevator and depressor groups. The collective term 'hamstrings' refers to four muscles- semimembranosus (SM), semitendinosus (ST), biceps femoris long head (BFlh) and biceps femoris short head (BFsh). The hamstring muscles are the major flexors of the knee and also aid hip extension. Trigger point is classically defined as a hyperirritable spot in the skeletal muscle that is associated with a hypersensitive palpable nodule in a taut band which is painful on compression and can give rise to characteristic referred pain, motor dysfunction, and autonomic phenomena. Latent trigger points located in the muscles can interfere with muscular movement patterns, cause cramps, and reduce muscle strength. Active MTrPs can be associated with a reduced range of motion through muscle dysfunction and muscle weakness, causing orefacial pain, MTrPs in the masticatory muscles may restrict active maximum mouth opening (MMO).

It is possible that stretching the hamstring muscles may activate the dorsal periaqueductal grey area of the midbrain [PAG], and activate descending inhibitory control pathways. It is known that descending projections from the PAG to the medulla have collateral branches that terminate in various areas including the upper cervical spinal cord. Convergence of the nociceptive afferents from the receptive fields of cervical roots C1-C3 and those of the trigeminal nerve, which include the masseter muscle, occurs in the nucleus caudalis. If hamstring muscle stretching is capable of activating the PAG, then decreased sensitivity should affect a greater number of muscles, including the remaining masticatory muscles.

Muscle energy technique (MET) is a manual technique developed by osteopaths that is now used in many different manual therapy professions. It is claimed to be effective for a variety of purposes, including lengthening a shortened or contractured muscle, strengthening muscles, as a lymphatic or venous pump to aid the drainage of fluid or blood, and increasing the range of motion (ROM) of a restricted joint. MET may influence pain mechanisms and promote hypoalgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 25 to 50 years..
2. Diagnosis of trps using the diagnostic criteria:

   * Presence of palpable taut band in a skeletal muscle.
   * Presence of hypersensitive tendor spot in a taut band
   * Spontaneous response of the typical referred pain pattern.
   * A local twitch response provided by snapping palpation of taut band.
   * Reproduction of the typical referred pain pattern of Trp in response to compression.
3. Reduced mouth opening < 40nm

Exclusion Criteria:

* Diagnosis of fibromyalgia.
* History of whiplash injury
* History of any surgery in the cranio cervical region
* Having under gone any myofacial pain therapy
* No lower extremity or low back pathology.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale VAS | 2 weeks
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.

SECONDARY OUTCOMES:
Inch Tape | 2 weeks
  A measuring tape is a flexible tool used for measuring. It is marked in centimeters and inches.
Jaw Functional Limitation Scale | 2 weeks
  The JFLS-20 is an organ-specific instrument comprising 3 constructs for assessing functional status of the masticatory system; the 3 scales exhibit properties that are ideal for both research and patient evaluation in patient groups with a range of functional limitations of the jaw.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No